CLINICAL TRIAL: NCT00104026
Title: Genes Associated With Hereditary and Drug-Induced Gingival Overgrowth
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050103; 05-D-0103
Record Dates: First submitted 2005-02-18; First posted 2005-02-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-19

CONDITIONS: Gingival Overgrowth
Keywords: Periodontal Disease; Dilantin; Cyclosporin; Calcium-Channel Blockers; Genetics; Hereditary Gingival Fibromatosis; HGF; Gingival Overgrowth; Gum Overgrowth
MeSH Terms: conditions — Gingival Overgrowth; Periodontal Diseases; Fibromatosis, Gingival, Hereditary

SUMMARY:
This study will examine common features of gingival overgrowth (excessive growth of the gums around the teeth) that develops in patients with the hereditary form of the condition and in those who develop the condition as a side effect of medications. A better understanding of gingival overgrowth may help scientists develop medications with fewer oral side effects.

Patients of any age with hereditary gingival fibromatosis and their blood relatives, and patients of any age with gingival overgrowth who are taking medications associated with development of the disorder, including phenytoin (diphenylhydantoin or Dilantin), cyclosporine, and calcium-channel blockers, may be eligible for this study.

Participants undergo a medical and dental history, including a history of medication use; detailed examination of the teeth, periodontium, head, and neck; photographs of teeth with gingival overgrowth; dental x-rays; and blood tests. DNA is extracted from a blood sample to look for genes related to gingival overgrowth.

Patients with gingival overgrowth are offered two options, as follows:

* Tissue biopsy: A tissue sample is taken from each affected site, with a maximum of three biopsies. For the procedure, lidocaine is first injected into the gum to numb the tissue. Then, a cookie-cutter instrument is pushed into the numbed skin, and a small piece of tissue is removed.
* Gingivectomy: Surgical removal of the overgrown gingival.

DETAILED DESCRIPTION:
The purpose of this protocol is twofold: 1) to continue identification of genes associated with hereditary gingival fibromatosis (HGF), a type of gingival overgrowth 2) to investigate the genes up-regulated by medications that induce gingival overgrowth. These studies will establish if common mechanisms are involved in the hereditary and drug-induced processes. If a common pathway is identified, it could lead to the development of assays that could be used to screen new medications for their potential deleterious effects on periodontal tissues. In addition, understanding the mechanisms involved in gingival overgrowth could lead to the development of tissue engineering approaches to repair gingival defects. Genes will be identified from DNA samples collected from patients with hereditary gingival fibromatosis. These will be compared with DNA and tissue samples taken from patients taking medications known to induce gingival overgrowth (phenytoin, cyclosporine and calcium channel blockers).

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients of any age, gender, and racial/ethnic group with hereditary gingival fibromatosis (HFG) as diagnosed with HGF by clinical appearance that consists of attached gingival covering the lower 1/3 or more of the clinical crowns of teeth in an individual not taking medications associated with gingival changes.

Blood relatives of affected individuals who are at risk of inheriting HGF.

Patients of any age, gender, and racial/ethnic group taking one of the three medications associated with drug-induced gingival overgrowth (phenytoin diphenylhydantoin or Dilantin, cyclosporine, or calcium-channel blockers).

Patients with six or more teeth.

EXCLUSION CRITERIA:

Patients with significant cognitive impairment.

Pregnant patients or lactating patients.

Patients unwilling to give informed consent.

Patients with less than six teeth.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-02-15; Study Completion 2011-04-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Boratynska M, Radwan-Oczko M, Falkiewicz K, Klinger M, Szyber P. Gingival overgrowth in kidney transplant recipients treated with cyclosporine and its relationship with chronic graft nephropathy. Transplant Proc. 2003 Sep;35(6):2238-40. doi: 10.1016/s0041-1345(03)00800-5. PMID 14529900
- [Background] Casetta I, Granieri E, Desidera M, Monetti VC, Tola MR, Paolino E, Govoni V, Calura G. Phenytoin-induced gingival overgrowth: a community-based cross-sectional study in Ferrara, Italy. Neuroepidemiology. 1997;16(6):296-303. doi: 10.1159/000109700. PMID 9430129
- [Background] Ellis JS, Seymour RA, Taylor JJ, Thomason JM. Prevalence of gingival overgrowth in transplant patients immunosuppressed with tacrolimus. J Clin Periodontol. 2004 Feb;31(2):126-31. doi: 10.1111/j.0303-6979.2004.00459.x. PMID 15016038